CLINICAL TRIAL: NCT07172971
Title: duCHennE caRdiomyopathy mItigation Sglt2 inHibitor
Brief Title: Sodium/Glucose Cotransporter-2 Inhibitors (SGLT2i) Therapy in Duchenne Cardiomyopathy
Acronym: CHERISH
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Larry W. Markham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Larry W. Markham, Professor of Pediatrics, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 28323; 1R61HL180327-01 (NIH)
Record Dates: First submitted 2025-08-07; First posted 2025-09-15 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: Cardiomyopathy; Heart failure; Muscular dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Cardiomyopathies; Heart Failure; Muscular Dystrophies | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dosing (Experimental): At the initial stage, investigators will allocate 3 subjects to 5 mg and 3 subjects 10 mg depending on their body weight (i.e., 5 mg for children with weight les than 40 kg, 10 mg for those with greater than 40 kg).
  Interventions: Drug: SGLT-2 inhibitor
- Pharmacokinetics (Experimental): In the second stage, based on the Pharmacokinetics (PK) analysis results from the initial 6 subjects divided in 5 mg and 10 mg dose groups, the next dose will be determined, for which the remaining 4 subjects will be allocated. The next dose decision will be made based on the target drug concentration levels along with the estimated PK parameters (e.g., the area under the drug concentration time curve and the maximum concentration), which correspond to adults PK and drug levels.
  Interventions: Drug: SGLT2 inhibitor

INTERVENTIONS:
Drug: SGLT-2 inhibitor — SGLT-2 inhibitor will be given once daily by mouth
  Arms: Dosing
Drug: SGLT2 inhibitor — SGLT-2 inhibitor will be given once daily by mouth
  Arms: Pharmacokinetics

SUMMARY:
This is a pharmacokinetic study (PK Study) to better understand empagliflozin dosing in pediatric Duchenne muscular dystrophy patients. Empagliflozin is currently used off-label in this population due to the mortality benefits seen in adult cardiomyopathy and heart failure. Investigators will perform PK studies in DMD patients of various ages and weights to better understand the PK profile (absorption, distribution, metabolism, excretion) and dosing to better treat Duchenne cardiomyopathy.

DETAILED DESCRIPTION:
Duchenne muscular dystrophy (DMD) is an X-linked skeletal and cardiac myopathy resulting from a defect in the gene coding for dystrophin. DMD myopathy leads to loss of ambulation, respiratory failure, cardiomyopathy (CM), and premature death. There is no cure, and while gene therapies now have approval, their cardiac effects are largely unstudied. Supportive care advances have decreased death from respiratory failure but have simultaneously unmasked the fully penetrant CM phenotype, which is now the leading cause of death in DMD.

Investigators have documented that DMD CM progresses from normal imaging to diastolic dysfunction with subtle strain abnormalities to manifest systolic dysfunction; these changes correspond pathologically with myocardial inflammation and progressive increase in myocardial fibrosis and fibrofatty infiltration. Large areas of fibrofatty replacement visible on cardiac magnetic resonance (CMR) are felt to be irreversible, meaning that for optimal benefit, therapy must begin before these changes have occurred. Guideline-directed medical therapy (GDMT) is increasingly applied in DMD CM care, but individual response to these therapies is suboptimal and often only serves to minimally delay the inevitable progression to heart failure and early death. There is a critical need for the application of new CM therapeutics in DMD.

Sodium/glucose cotransporter-2 inhibitors (SGLT2i) have resulted in mortality benefits in adult CM. The mechanism of this beneficial effect is unknown, but several factors translating to DMD suggest that SGLT2i could have potential for DMD CM: 1) improved cardiac energetics and metabolism; 2) improved mitochondrial function and reduced oxidative stress; 3) reduction in inflammation; 4) inhibition of myocardial fibrosis; 5) reduction in sarcoplasmic calcium leak; 6) improved sympathetic overdrive. While the use of SGLT2i in pediatric patients with significant LV dysfunction has become more common, there are many significant unanswered questions. PK data are limited, and many patients are dosed based on glucosuria, which is not a proven method to determine efficacy or exclude side-effects. The potential for earlier therapy in DMD, before irreversible changes, is immense; however, an understanding of appropriate dosing for children with DMD is necessary before this can be achieved.

ELIGIBILITY:
Inclusion Criteria:

* Clinical phenotype of DMD confirmed with muscle biopsy or genotype
* Presence of late gadolinium enhancement (LGE) imaging by CMR
* Either normal or mildly depressed systolic function (LVEF>40%)
* ≥8 years old and ≤18 years old

Exclusion Criteria:

* Current investigational therapy that may affect cardiovascular function

  * Additional genetic or congenital abnormality that may affect cardiovascular function or progression
  * Contraindication to or inability to undergo CMR
  * Symptomatic heart failure
  * History of ketoacidosis or hypersensitivity to SGLT2i therapy
  * Type 1 diabetes
  * Renal disease or history of frequent urinary tract infections or genitourinary skin infections

Ages: 8 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Male
Enrollment: 10 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Medication dose | From enrollment to 12 month analysis
  DMD patients will be given different doses of medication to better understand the most appropriate dosing of medication in this rare disease population. Because age and weight can impact how a DMD patient absorbs and metabolizes medication, the study will include DMD patients of various ages and weights. This includes giving a dose of medication and measuring drug levels in blood over a 24 hour period of time.

SECONDARY OUTCOMES:
Medication absorption in blood | Enrollment to 12 month analysis
  DMD patients will be given different doses of medication to better understand the most appropriate dosing of medication in this rare disease population. Because age and weight can impact how a DMD patient absorbs medication, the study will include DMD patients of various ages and weights. This includes giving a dose of medication and measuring drug levels in blood over a 24 hour period of time.
Medication Excretion or Elimination from blood | Enrollment to 12 months
  DMD patients will be given different doses of medication to better understand the most appropriate dosing of medication in this rare disease population. Because age and weight can impact how a DMD patient absorbs and excretes or eliminates a medication, the study will include DMD patients of various ages and weights. This includes giving a dose of medication and measuring drug levels in blood over a 24 hour period of time.

CONTACTS AND LOCATIONS:
Overall Officials: Larry W. Markham, MD, Principal Investigator — Riley Children's Hospital
Locations (1):
- Riley Hospital at Indiana University Health, Indianapolis, Indiana, United States